CLINICAL TRIAL: NCT00713791
Title: A Phase I, Randomised, Single-blind, Single-centre, Incomplete-block Crossover, Relative Bioavailability Study in Healthy Male Subjects for ZD4054 (Zibotentan) Immediate Release Tablets
Brief Title: Relative Bioavailability Study in Healthy Male Subjects for ZD4054 (Zibotentan) Immediate Release Tablets.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Thomas Morris, Medical Science Director, AstraZeneca, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: D4320C00029; ZD4054IL0029
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Healthy Volunteers; ZD4054
MeSH Terms: interventions — ZD4054

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- 1 (Experimental): There are 5 variations of the ZD4054 (Zibotentan) 10mg tablet - A, B, C, D, and E. A minimum washout period of 1 week will occur between each treatment period.
  Interventions: Drug: ZD4054

INTERVENTIONS:
Drug: ZD4054 — Treatment period 1: 10mg oral solution
  Other Names: Zibotentan
Drug: ZD4054 — Treatment period 2: 3 of the 5 tablet variations (A-E) to be taken in a random sequence, but not the same tablet twice.
  Other Names: Zibotentan
Drug: ZD4054 — Treatment period 3: 3 of the 5 tablet variations (A-E) to be taken in a random sequence, but not the same tablet twice.
  Other Names: Zibotentan
Drug: ZD4054 — Treatment period 4: 3 of the 5 tablet variations (A-E) to be taken in a random sequence, but not the same tablet twice.
  Other Names: Zibotentan

SUMMARY:
This study is designed to see how different formulations of ZD4054 (Zibotentan) are absorbed by the body. As for all clinical trials, safety and tolerability of the drug will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Normal resting 12-lead ECG with normal QTc interval (<450 msec)
* Negative screens for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV) at screening

Exclusion Criteria:

* Receipt of another new chemical entity in the 4 months before dosing in this study; participation in another study and participation in a non-invasive methodology study in which no drugs were given within 30 days before dosing in this study
* Risk (in the investigator's opinion) of transmitting, through blood or other body fluids, the agents responsible for acquired immune deficiency syndrome (AIDS), hepatitis B or hepatitis C
* Judgement by the investigator, that the healthy volunteer should not participate in the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-06; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
characterise and compare the plasma concentration-time profiles for ZD4054 (Zibotentan) when administered as reference oral solution formulation and as 5 solid oral formulations. | 00.50mins, 01.00, 01.15, 01.30, 01.45, 02.00, 02.30, 03.00, 04.00, 06.00, 08.00, 12.00, 24.00, 36.00, 48.00, 72.00, 96.00hrs

SECONDARY OUTCOMES:
characterise and compare pharmacokinetic parameters for ZD4054 (Zibotentan) when administered as an oral solution and as 5 solid oral formulations and to assure the safety of all healthy volunteers by assessment of vital signs, ECG, Labs, and AEs | 00.05, 00.10, 00.15, 00.20, 00.30, 00.40, 00.50mins, 01.00, 01.15, 01.30, 01.45, 02.00, 02.30, 03.00, 04.00, 06.00, 08.00, 12.00, 24.00, 36.00, 48.00, 72.00, 96.00hrs
To assure the safety of all subjects by assessment of vital signs, ECG, clinical chemistry, haematology, urinalysis and adverse events. | From time of Consent to Last Visit

CONTACTS AND LOCATIONS:
Overall Officials: Sylvan Hurewitz, Principal Investigator — AZ Clinical Pharmacology Unit, Philadelphia, USA
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States